CLINICAL TRIAL: NCT01713387
Title: A Phase I Study of Adjuvant Chemotherapy With Gemcitabine Plus S-1 in Patients With Biliary Tract Cancer Undergoing Curative Resection Without Major Hepatectomy
Brief Title: A Phase I Study of Adjuvant Chemotherapy With GS in Biliary Tract Cancer Undergoing Resection Without Major Hepatectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kansai Hepatobiliary Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KHBO1202; UMIN000007454 (Registry Identifier: UMIN)
Record Dates: First submitted 2012-09-18; First posted 2012-10-24 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-08

CONDITIONS: Biliary Tract Cancer
Keywords: adjuvant chemotherapy
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gemcitabine , S-1 (Experimental): Level-2 Gem 800mg/msq, S-1 50mg/msq Level-1 Gem 800mg/msq, S-1 65mg/msq Level 1 Gem 1000mg/msq, S-1 65mg/msq Level 2 Gem 800mg/msq, S-1 80mg/msq
  Interventions: Drug: Gemcitabine, S-1

INTERVENTIONS:
Drug: Gemcitabine, S-1 — Dose of gemcitabine and S-1 and treatment schedule
  Other Names: Gemcitabine;gemzer , S-1;TS-1

SUMMARY:
To decide maximum tolerated dose and recommended dose of treatment using gemcitabine plus S-1 combination therapy in patients with biliary tract cancer undergoing resection without major hepatectomy

DETAILED DESCRIPTION:
Surgery currently remains the only potentially curative treatment for biliary tract cancer (BTC), and most patients develop recurrence. Therefore, effective adjuvant chemotherapy is required to increase the curability of surgery and to prolong the survival in these patients. However, to date, no standard adjuvant chemotherapy has been established, and a guideline for BTC treatment recommends that trials of adjuvant chemotherapy be carried out.

Recently, there are two reports about gemcitabine (GEM) + S-1 combination (GS)chemotherapy after surgical resection for patients with BTC. At Iwate Medical University, Takahara, et al., performed a phase I study using a regimen of repeating 28 days as 1 course. Patients received GEM on day 1 and day 15, and S-1 from day 1 to day 14. The recommended dose is 1,000 mg/m² of GEM and S-1 80 mg/m² after a pancreatoduodenectomy. The 2-year survival rate of the 34 patients that received the GS therapy was 78.6% (Cancer Chemother Pharmacol. 2012 May;69(5):1127-33). At Hiroshima University, a cycle of chemotherapy consisted of intravenous GEM of 700 mg/m² on day 1 and oral S-1 of 50 mg/m² for 7 consecutive days, followed by a 1-week break from chemotherapy (14days as 1 course). Fifty patients received GS therapy and had a significantly better 3-year survival rate (57%) compared with 53 cases of surgery alone (30%). The GS adjuvant chemotherapy was feasible and the adverse event was minimal (Ann Surg. 2009 Dec;250(6):950-6).

Thus, the regimens of these two studies were 14 or 28 days as 1 course. There was no regimen that consisted of GEM on day 1, 8 and S-1 for 14 consecutive days, followed by a 1-week break from chemotherapy (21days as 1 course), which is frequently used for unresectable BTC and pancreatic cancer.

Though a hepatectomy is frequently performed during surgery for BTC, it is unclear if the effect of the anticancer agent is affected by a hepatectomy. Because GEM is metabolized by cytidine deaminase primarily in the liver, the ability to metabolize GEM after a hepatectomy is thought to decrease. Some clinical studies demonstrated that patients who had undergone a hepatectomy could not tolerate the standard dose and schedule of GEM. For adjuvant chemotherapy with GEM, it is necessary to separately examine whether or not the patient has undergone a hepatectomy.

Considering these present conditions, we aimed to assess the safety and efficacy of GEM + S-1 combination chemotherapy (21days as 1 course regimen, which is frequently used for unresectable BTC) for BTC with the patients undergoing curative resection without a hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Biliary tract cancer (BTC) with more than stage IB
2. BTC undergoing R0 or R1 resection without major hepatectomy
3. Older than 20 years old
4. PS 0 or 1
5. No treatment other than surgery
6. No dysfunction of main organs
7. Possible oral intake
8. Treatment start; after 4 weeks and within 12 weeks after surgery
9. Obtained written informed consent

Exclusion Criteria:

1. Patients with resection of major hepatectomy
2. Patients with double cancers
3. Patients having severe allergy
4. Patients with severe organ dysfunction
5. Patients with active infectious disease
6. Pregnancy
7. Patients with severe psychological disease
8. Patients seem inadequate for this study by investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 6 weeks
  To establish the maximum tolerated dose of gemcitabine plus S-1 in patients with biliary tract cancer undergoing curative resection without major hepatectomy

SECONDARY OUTCOMES:
Number of Participants with dose limiting toxicity | At the end of adjuvant chemotherapy (6 months)
  Dose limiting toxicity is defined as follows
  1. Grade 4 neutropenia, thrombocytopenia
  2. Grade 3 or 4 febrile neutropenia
  3. Grade 3 or 4 non-hematological adverse events unless unresponsive to treatment
  4. Any adverse events resulting in interruption of dosing on day 8 in both the two courses
  5. Any adverse events resulting in dose modification or delay of longer than 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hideyoshi Toyokawa, MD, PhD, Study Director — Kansai Medical University
Locations (1):
- Kansai Medical University, Hirakata, Osaka, Japan